CLINICAL TRIAL: NCT01454856
Title: Perioperative Evaluation of Immuno-inflammatory Parameters
Status: Terminated | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Forget Patrice, Principal Investigator, Université Catholique de Louvain
Other Study IDs: 2011/30MAI/218
Record Dates: First submitted 2011-10-05; First posted 2011-10-19 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Combined Inflammatory and Immunologic Defect
MeSH Terms: conditions — Combined Inflammatory and Immunologic Defect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and cells (PBMCs) frozen in cryotubes
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Surgical cancer patients: No modification of the treatment
- Non-surgical cancer patients: No modification of the treatment
- Surgical non-cancer patients: No modification of the treatment
- Non-surgical non-cancer patients: No modification of the treatment

SUMMARY:
This study consists of evaluations, using blood tests, various immune, inflammatory and coagulation parameters in the perioperative settings (different substudies), without changing anything to what is expected.

This will allow us to clarify the possible impact of surgery and analgesia on perioperative activation of these pathways.

DETAILED DESCRIPTION:
A significant number of published data can be concluded that surgery and anesthetic and analgesic techniques have an impact on immunity and inflammation.

However, none of these studies have been performed with modern techniques, much more reliable evaluation of immune activity, such as the assessment of monocytic degranulation by flow cytometry.

It is therefore important to document immune activity using these new techniques, our patients, perioperative. This will be analyzed, so observational, the potential impact of different therapeutic interventions the patient receives.

This study consists of evaluations, using blood tests, various immune, inflammatory and coagulation parameters in the perioperative settings (different substudies), without changing anything to what is expected.

This will allow us to clarify the possible impact of surgery and analgesia on perioperative activation of these pathways.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients (and controls)

Exclusion Criteria:

* Immune disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of patients
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Immune parameters (immunocytes phenotype) | baseline up to 8 days (return to baseline)
  Function tests and surface markers

SECONDARY OUTCOMES:
Long term outcome | 5 years
  General morbidity and mortality
Coagulation parameters (like platelet function) (substudy) | perioperative period (up to 3 days)
  Function tests and surface markers
Inflammatory markers (cytokines) (substudy) | baseline up to 8 days (return to baseline)
  Intracellular FACS and ELISA measures

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Forget, M.D., Principal Investigator — UCL
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium